CLINICAL TRIAL: NCT00796237
Title: Effects of Whole Body Vibration Training on Bone Health, Physical Fitness, and Neuromotor Performance in Individuals With Subacute Stroke: a Randomized Controlled Trial
Brief Title: Effects of Whole Body Vibration in Subacute Stroke Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Hong Kong Polytechnic University (Other)
Collaborators: Tung Wah Hospital (Other)
Responsible Party: Marco Yiu-Chung Pang, Hong Kong Polytechnic University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UW-08-032
Record Dates: First submitted 2008-11-21; First posted 2008-11-24 (Estimated); Last update posted 2011-08-09 (Estimated); Status verified 2011-08

CONDITIONS: Stroke
Keywords: stroke; bone; gait; muscle; vibration; motor balance
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- WBV (Experimental): In their regular physiotherapy sessions, the subjects in the experimental group will receive whole body vibration therapy for a duration of 4 weeks during their stay in the Tung Wah Hospital.
  Interventions: Device: Whole body vibration therapy
- CON (Active Comparator): The subjects in this group will not receive whole body vibration therapy.
  Interventions: Other: standing on the vibration platform but no vibration will be applied

INTERVENTIONS:
Device: Whole body vibration therapy — In their regular physiotherapy sessions, the subjects in the experimental group will receive WBV (20-240Hz, 10-minute sessions, 1 session per day, 5 sessions per week). The vibration loading will be carried out using the Fit-Vibe System (Germany), which is a vibration platform that is capable of generating vertical vibration.
  Arms: WBV
Other: standing on the vibration platform but no vibration will be applied — The subjects in this group will perform the same exercises on the vibration platform as in the experimental group for the same duration, but no vibration will be given.
  Arms: CON

SUMMARY:
The overall aim of the proposed study is to determine whether whole body vibration is beneficial in promoting bone turnover, physical fitness and neuromotor performance in patients with subacute stroke.

DETAILED DESCRIPTION:
Brief periods of Whole body vibration (WBV) have been shown to improve bone density in post-menopausal women and children with cerebral palsy. In addition to the apparent benefits on bone health, WBV has been shown to increase muscle strength, postural control, muscular blood flow and oxygen uptake in various populations. Therefore, WBV can potentially be used as a tool to improve muscle strength, balance, and cardiovascular performance, especially for those with relatively low level of functioning. Stroke patients are therefore possible beneficiaries of WBV, as they often demonstrate muscle weakness, balance deficits, and poor cardiovascular function, in addition to bone loss. Only one pilot study has examined the effects of WBV in stroke patients. Van Nes et al.showed that postural stability in chronic stroke patients is improved after a few minutes of WBV at 30Hz and 3mm amplitude. The overall aim of the proposed study is to determine whether whole body vibration is beneficial in promoting bone turnover, physical fitness and neuromotor performance in patients with subacute stroke.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of stroke
* medically stable
* able to understand simple verbal commands
* of chinese origin

Exclusion Criteria:

* previous stroke in addition to the current admission
* other neurological conditions, in addition to stroke
* significant musculoskeletal or vascular conditions in the lower extremity
* metal implants in the lower extremity
* previous fracture in the lower extremity
* are taking or were taking bone resorption inhibitors

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2008-05; Primary Completion 2011-12 (Estimated); Study Completion 2011-12 (Estimated)

PRIMARY OUTCOMES:
Level of bone resorption marker CTx | baseline, immediately after treatment, and 2-month follow-up
Level of bone formation marker, BSAP | baseline, immediately after treatment, and 2-month follow-up

SECONDARY OUTCOMES:
Six minute walk test | baseline, immediately after treatment, and 2-month follow-up
Ankle arm index | baseline, immediately after treatment, and 2-month follow-up
Functional Ambulation category | baseline, immediately after treatment, and 2-month follow-up
Leg muscle strength (hand-held dynamometry) | baseline, immediately after treatment, and 2-month follow-up
Berg Balance Scale | baseline, immediately after treatment, and 2-month follow-up
Modified Ashworth Scale of Spasticity | baseline, immediately after treatment, and 2-month follow-up
Sensory threshold to light touch in the foot | baseline, immediately after treatment, and 2-month follow-up
Fugl-Meyer Motor Assessment | baseline, immediately after treatment, and 2-month follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Marco YC Pang, PhD, Principal Investigator — The Hong Kong Polytechnic University
Locations (1):
- Tung Wah Hospital, Hong Kong, Hong Kong

REFERENCES:
- [Background] Bogaerts A, Delecluse C, Claessens AL, Coudyzer W, Boonen S, Verschueren SM. Impact of whole-body vibration training versus fitness training on muscle strength and muscle mass in older men: a 1-year randomized controlled trial. J Gerontol A Biol Sci Med Sci. 2007 Jun;62(6):630-5. doi: 10.1093/gerona/62.6.630. PMID 17595419
- [Background] Verschueren SM, Roelants M, Delecluse C, Swinnen S, Vanderschueren D, Boonen S. Effect of 6-month whole body vibration training on hip density, muscle strength, and postural control in postmenopausal women: a randomized controlled pilot study. J Bone Miner Res. 2004 Mar;19(3):352-9. doi: 10.1359/JBMR.0301245. Epub 2003 Dec 22. PMID 15040822
- [Background] van Nes IJ, Geurts AC, Hendricks HT, Duysens J. Short-term effects of whole-body vibration on postural control in unilateral chronic stroke patients: preliminary evidence. Am J Phys Med Rehabil. 2004 Nov;83(11):867-73. doi: 10.1097/01.phm.0000140801.23135.09. PMID 15502741
- [Background] Torvinen S, Kannus P, Sievanen H, Jarvinen TA, Pasanen M, Kontulainen S, Nenonen A, Jarvinen TL, Paakkala T, Jarvinen M, Vuori I. Effect of 8-month vertical whole body vibration on bone, muscle performance, and body balance: a randomized controlled study. J Bone Miner Res. 2003 May;18(5):876-84. doi: 10.1359/jbmr.2003.18.5.876. PMID 12733727
- [Background] Ward K, Alsop C, Caulton J, Rubin C, Adams J, Mughal Z. Low magnitude mechanical loading is osteogenic in children with disabling conditions. J Bone Miner Res. 2004 Mar;19(3):360-9. doi: 10.1359/JBMR.040129. Epub 2004 Jan 27. PMID 15040823